CLINICAL TRIAL: NCT05589428
Title: Effectiveness of Low-salt Bread on the Total Sodium Intake in Patients With Chronic Heart Failure and Chronic Kidney Disease (LoSa Pilot Study)
Brief Title: Low-salt Bread in Heart Failure, Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VieCuri Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: NL47820.068.14; NL47820.068.14 (Other: ToetsingOnline ID/CCMO ID); 47820.068.14 (Other: METc)
Record Dates: First submitted 2022-05-03; First posted 2022-10-21 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure, Systolic; Sodium Imbalance; Food Selection
MeSH Terms: conditions — Heart Failure, Systolic; Food Preferences

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal bread
  Interventions: Other: Placebo
- Low sodium bread (Experimental): Low sodium bread
  Interventions: Dietary Supplement: Low sodium bread

INTERVENTIONS:
Dietary Supplement: Low sodium bread — Bread low in sodium
  Arms: Low sodium bread
Other: Placebo — Normal bread from bakery
  Arms: Placebo

SUMMARY:
SUMMARY Rationale Patients with heart failure may suffer from a poor quality of life (QoL) due to frequent hospital admittance, medication intake, and symptoms as a result of progression of their disease. The general salt intake in the Dutch population is too high, leading indirectly to hypertension resulting in worsening of cardiovascular disease such as heart failure. Patients with heart failure are highly salt sensitive. A quarter of the daily salt intake originates from bread. Salt restriction is difficult to maintain.

The aim of this study is to lower the daily salt intake by providing a palatable low salt bread to patients with heart failure. This may lead to a stable disease and therefore an improvement in quality of life.

Objective The aim of this study is to investigate whether substitution of normal bread by a new palatable form of low salt bread is effective in reducing salt intake in patients with chronic heart failure. The investigators will evaluate the effectiveness, the compliance and the outcome of the presumed salt reduction.

Study design This is a single center, randomized, double blinded, cross-over trial with a follow-up period of twelve weeks performed in VieCuri, Medical Centre in Venlo.

Study population In this study, 20 patients visiting the outpatient clinic with heart failure NYHA class 3-4 will be included. All patients are 18 years or older.

Intervention Given the study design all 20 patients receive a low salt bread (0.05 gram sodium per slice) for one period and received bread with a normal amount of sodium (0.35 gram sodium per slice) in the other period. After six weeks follow up, the groups change the intervention.

Main study parameters/endpoints The investigators expect a reduction of daily salt intake of 1.5 gram sodium by an average of 5 slices bread a day.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness Patients should visit the hospital three times. Prior the hospital visit they have to collect 24- hour urine. During all visits blood samples will be taken and a physical exam is performed. Also blood pressure will be measured. Most of these parameters are also collected for clinical purposes. Patients should at the same time report their daily intake in a personal food diary and fill in questionnaires about their opinion of the bread and quality of life.

DETAILED DESCRIPTION:
The study population is randomized and participants are chosen based on the diagnosis of chronic heart failure. After participants were informed and consented by telephone and in writing, secondary data were collected (primary etiology of disease, age, height, weight, BMI, medication). Patients were randomized and the study bread was prepared by a baker. Only the baker was aware of which bread was the normal bread and which was the study bread. Both loaves were labeled. Participants, investigators and outcome assessors were blinded to the assignment.

The study was a crossover study. The participants were followed for a period of 12 weeks, during which they took 6 weeks of low-salt bread and 6 weeks of normal bread. A minimum intake of 4-5 slices of bread per day was requested for participation in the study. Two different loaves were made; a loaf with 0.35 grams of salt per slice of bread (normal) and a loaf with 0.05 grams of salt per slice of bread (low salt content). Based on an average bread intake of 4-5 slices per day, a clinically relevant difference in sodium excretion between the interventions of 1.2-1.5 grams per day was expected. Patients were informed by telephone and in writing about the need to eat at least 4 slices of bread per day. It was expressly stated that if the patient could not achieve this, participation was not possible.

These intervention groups are thus as follows:

* Group 1: starts with the Scelta bread with a normal amount of sodium (0.4 grams sodium per slice)
* Group 2: starts with the low sodium Scelta bread (0.1 gram sodium per slice). During this period, the subjects kept a food diary 1 day per week (12 days in total).

At three different times there were contact moments (45 minutes) with the patient and data were collected consisting of: 15 minutes blood pressure measurement, collection of 24-hour urine, body weight and bioimpedance measurement, a short physical examination, filling in questionnaire about quality of life and nutrition and finally a blood test. The included patients were also seen by the dietitian immediately after contact with the researcher. They also received dietary advice regarding salt restriction.

Inclusion criteria

Patients may participate if they meet the following criteria:

* Age over 18 years
* Heart failure NYHA class III-IV or LVEF < 35%, in a stable condition (no medication changes in the past two weeks)
* Being able to issue written informed consent
* Dutch speaking and reading

Exclusion criteria

Patients may not participate in the study if they meet the following criteria:

* Pregnancy or breastfeeding
* Participate in another study during the intervention
* Hyponatraemia < 130 mmol/L
* Hypokalaemia < 3.4 mmol/l
* Hyperkaliemia > 5.5 mmol/l
* Cognitive Impairment
* Blood pressure systolic below 100 mmHg or diastolic below 50 mmHg
* Allergic reaction to mushrooms, silica, corn and gluten
* Life expectancy shorter than one year.

Variables Primary variable The primary endpoint of this study is the reduction of salt intake. This is assessed with the oral intake of salt, which will be determined using a food diary kept by the participant. The participant's compliance can also be viewed here. This is compared to the amount of sodium in the urine. It is hypothesized that the use of low-salt bread leads to a reduction in total daily salt intake, resulting in decreased urinary sodium excretion.

Secondary Variables

The secondary variables are:

* Blood pressure
* Weight
* Body composition and fluid status (intra and extra cellular) by means of a Body Composition Monitor (BCM measurement)
* Venous blood: sodium, BNP
* Symptoms of heart failure according to the Minnesota Living with Heart Failure questionnaire
* Taste of bread

Data collection The diet of the participants was examined together with the dietician on the first outpatient visit. Any details were discussed immediately and advice followed if necessary. The patients all kept a food diary in which they wrote down all oral intake one day a week. They were also asked to record the oral intake the day before the outpatient visit. In this way the dietitian could calculate the salt intake and this could be compared with the sodium in the urine.

Blood pressure was measured three times over a period of 15 minutes. The last measured blood pressure was used in the analysis.

The fluid balance (intra and extra cellular volume) was measured using a Body Composition Monitor (BCM measurement) from Fresenius Medical care. This is a bioimpedance spectroscopy device for clinical use, validated with isotope dilution methods. The 'overhydration' parameter was used for the follow-up. Overhydration represents the excess fluid that is almost exclusively stored in a patient's extracellular volume and is therefore part of the 'extracellular water' (ECW).

Labs were taken from patients during each outpatient visit. Several determinations were made for this. In order to answer the question, the BNP and sodium were considered the most important in this study. The biologically active B-type natriuretic peptide or brain natriuretic peptide (BNP) and the biologically inactive N-terminal proBNP (NT-proBNP) are substances produced by the heart that are released into the circulation and mainly provide information about the filling pressures of the heart . The accuracy of BNP plasma levels for the diagnosis of heart failure is comparable to that of NT-proBNP plasma levels.

The Minnesota Living with Heart Failure questionnaire was designed in 1984 to measure the effects of heart failure and heart failure treatments on an individual's quality of life. The content of the questionnaire was chosen to be representative of the ways in which heart failure can affect key physical, emotional, social and mental dimensions of quality of life. The list has been developed for use in daily practice. To measure the effects of symptoms, functional limitations, and psychological stress of heart failure on quality of life, the MLHFQ asks each person to rate, using a 6-point (zero to five) scale, how much each of its 21 facets interferes with them. in daily life. The questionnaire assesses the impact of frequent physical symptoms such as shortness of breath, fatigue, peripheral edema and difficulty sleeping - and psychological symptoms of anxiety and depression. In addition, the effects of heart failure on physical and social functioning are also included in the measuring instrument. Because treatments may have side effects in addition to the symptoms and functional limitations of heart failure, questions about drug side effects, hospital stays, and costs of care were also included to help measure the overall impact of treatment on quality of life. Although the MLHFQ contains relevant aspects of the main dimensions of quality of life, the questionnaire was not designed to measure any particular dimension in isolation. The total score is presented in mean SD. The intervention group is compared with the control group. The NYHA classification is also reviewed with every outpatient check.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years;
* CHF NYHA III-IV or LVEF <35%, stable condition on optimal medical therapy: no medication changes in last two weeks prior to start study.
* Written informed consent
* Speak and read Dutch

Exclusion Criteria:

* Pregnancy or breastfeeding
* Participating in any other interventional research study during the same period
* Hyponatremia; sodium < 130 mmol/L
* Hypokaliemia < 3.4 mmol/l
* Hyperkaliemia > 5.5 mmol/l
* Cognitive impairment
* Blood pressure systolic below 100 mmHg OR diastolic below 50 mmHg
* Allergic reaction to mushrooms, silica, corn and gluten
* Life expectancy shorter than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Sodium excretion urine | 6 weeks
  24-hour urine sample will be analysed on sodium excretion. This will be measured at baseline and after each 6 week period.
  Also sodium, protein, albumin and creatinine concentration will be measured.

SECONDARY OUTCOMES:
Blood samples | 6 weeks
  the effect of the presumed lower salt intake, blood samples will be taken to measure sodium, potassium, creatinine and NT-proBNP. This will be measured at baseline and after each 6 week period.
Sodium intake | 12 weeks.
  Subjects are asked to fill in a personal food diary. One day a week for 12 weeks. Sodium intake will be measured'.
Taste of bread | 6 weeks
  During visits patients are asked about taste of bread via a questionnaire
Quality of Life Questionnaire | 6 weeks
  During visits patients are asked about QOL via a questionnaire
Blood pressure | 6 weeks
  During visits blood pressure will be measured non-invasively for 15 minutes. at baseline and at the end of each intervention
Body composition measurement with bioimpedance spectroscopy (BIS) | 6 weeks
  During visits excess fluid state (in Liters) will be measured non-invasively by applying the BCM Fresenius.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Meeder, MD PhD, Principal Investigator — VieCuri Medical Centre
Locations (1):
- ViecuriMC, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No